CLINICAL TRIAL: NCT05336045
Title: Satisfaction and Recovery After Trigger Finger Release- a Prospective Cohort Study With Weekly PROMs
Brief Title: Satisfaction and Recovery After Trigger Finger Release
Acronym: TH III
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Stromberg, senior consultant surgeon, MD, PhD, Sahlgrenska University Hospital
Other Study IDs: TriggerHappy III
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2023-11

CONDITIONS: Trigger Finger Disorder
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: trigger finger release — The A1 pulley and tendon sheath is divided in local anaestethic through a small incision in the palm

SUMMARY:
Trigger finger release is one of the most common procedures in hand surgery. However, little is known about the patient perceived outcome directly after surgery and the timespan to recovery of normal hand function.This study focuses on patient reported outcome scores within the first six weeks after surgery.

DETAILED DESCRIPTION:
Patients scheduled for release of trigger finger are assessed regarding the following outcome measures:

1. VAS score for pain
2. VAS score for finger movement
3. VAS score for fréquence of triggering
4. HAKIR questionnaire (validated instrument for hand function in the Swedish national hand registry)
5. Quick-DASH questionnaire.

After surgery, the patients records the following outcomes:

Each day: 1,2,3 and records of pain medication details Each week: 4,5

for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Trigger phenomenon and/or
2. Tenderness volarly to MCP joint of affected finger/thumb
3. Patient scheduled for trigger finger release
4. Signed informed consent

Exclusion Criteria:

1. Concomitant hand injuries/ conditions
2. Multiple fingers/thumbs to be treated
3. Unable to read/understand instructions in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for trigger finger release
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Self-assessed hand function | every week for 6 weeks
  change in total score of hand-specific questionnaire (HAKIR) week by week. Best score 100, worst 0

SECONDARY OUTCOMES:
Pain (assessed by patient) | 6 weeks
  change in Visual Analouge Scale-score day by day (0= worst, 10=best)
Movement of finger (self-assessed by patient) | 6 weeks
  change in Visual Analouge Scale-score day by day (0= worst, 10=best)
Frequency of trigger phenomenon (self-assessed by patient) | 6 weeks
  change in Visual Analouge Scale-score day by day (0= worst, 10=best)

CONTACTS AND LOCATIONS:
Locations (1):
- Alingsås lasarett, Alingsås, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
open repositry